CLINICAL TRIAL: NCT05069064
Title: Effect of Music on Pain and Satisfaction in Infertile Patients Undergoing Hysterosalpingography: a Randomized Controlled Trial
Brief Title: Effect of Music on Pain and Satisfaction in Infertile Patients Undergoing Hysterosalpingography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Collaborators: Hospital El Gezeera (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, assistant professor of obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: hysterosalpingography music
Record Dates: First submitted 2021-09-25; First posted 2021-10-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Hysterosalpingography
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- music group (Experimental): In the music group, music chosen by the participant will be played through a speaker by the nursing staff during outpatient hysteroscopy. Music will be played through a speaker instead of headphones in order to maintain good communication and interaction between the participant and the doctor.
  Interventions: Other: music
- non-music group (Other): Participants in the non-music group will undergo hysterosalpingography in the same setting and standard procedure without listening to any music.
  Interventions: Other: no music

INTERVENTIONS:
Other: music — In the music group, music that chosen by the participant will be played through a speaker by the nursing staff during outpatient hysteroscopy. Music will be played through a speaker instead of headphone in order to maintain a good communication and interaction between the participant and the doctor.
  Arms: music group
Other: no music — Participants in the non-music group will undergo hysterosalpingography in the same setting and standard procedure without listening to any music.
  Arms: non-music group

SUMMARY:
The aim of this study is to demonstrate the value of music in infertile patients undergoing hysterosalpingography on patients' level of pain and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Infertility; patients aged 19 to 42 years; candidate for hysterosalpingography.

Exclusion Criteria:

* Severe dysmenorrhea; pelvic infections; drug sensitivity; unwillingness to participate in the study; presence of psychiatric disorders, use of psychotropic medications; secondary infertility.

Ages: 19 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2021-10-05 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-15 (Estimated)

PRIMARY OUTCOMES:
pain During contrast medium injection | 5 minutes
  pain will be assessed by visual analog scale from 0 to 10

SECONDARY OUTCOMES:
pain after hysterosalpingography | 10 minutes
  pain will be assessed by visual analog scale from 0 to 10